CLINICAL TRIAL: NCT02196116
Title: Amyloïd Load in Elderly Population: Effect of Cognitive Reserve
Acronym: EDUMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation Plan Alzheimer (Other); General Electric (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CHUBX 2013/02
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Plaque, Amyloid; Cognitive Deficits
Keywords: Alzheimer disease; amyloid load; educational level; cognitive performances
MeSH Terms: conditions — Plaque, Amyloid; Cognition Disorders; Alzheimer Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Controls
  Interventions: Other: PET; Other: MRI; Other: neuropsychological tests
- Group 2 (Experimental): Cognitively-impaired subjects without dementia and without memory
  Interventions: Other: PET; Other: MRI; Other: neuropsychological tests
- Group 3 (Experimental): Cognitively-impaired subjects without dementia and with memory
  Interventions: Other: PET; Other: MRI; Other: neuropsychological tests

INTERVENTIONS:
Other: PET — PET Scan with [18F]-Flutemetamol
Other: MRI
Other: neuropsychological tests

SUMMARY:
This research aim to explore relationships between the presence of amyloid burden and cognitive performance, and its modulation by educational level. For this purpose we will combine Positron emission tomography (PET) imaging and neuropsychological assessment acquired on 3 groups of subjects, from two population-based cohorts "3C" and "AMIMage" The first group includes cognitively intact participants who will serve as controls, the second group, subjects with mild cognitive impairments without memory complaint and the third, subjects with both mild cognitive impairments and memory complaint.

DETAILED DESCRIPTION:
Influence of educational level on the relationship between disease-specific lesion development and cognitive function will be assessed, as measured by amyloid PET imaging and a battery of neuropsychological tests at the very early stages of the disease, comparatively to age-matched controls. In addition, this project will explore the influence of cognitive complaint.

It's assumed that 1) the amyloid-PET measures in age-matched controls and subjects from the two cohorts will correlate with cognitive performances; 2) the amyloid burden will be higher in high- than in low-educated subjects with similar cognitive impairment; and 3) similarly the amyloid burden will be higher in subjects with cognitive complaint compared to subjects without cognitive complaint.

Considering a longer term, the clinical follow-up of study participants will allow to investigate the prognosis value of amyloid load for improving the prediction of cognitive decline and disease progression.

ELIGIBILITY:
Inclusion Criteria:

Participation in the AMI or 3C cohorts Group 1- Controls

* MMSE > 24 or > 26 for low and high levels of education, respectively.
* Without memory impairment (for episodic memory) on the Free and Cued Selective Reminding Test RL/RI-16 items (FCSRT), free recall > 22 and total recall >42, according to the thresholds for population-based studies
* Without memory complaint
* Without dementia Group 2- Cognitively-impaired subjects without dementia and without memory complaints
* Mini Mental State Evaluation (MMSE) < 24 or < 26 for low and high levels of education, respectively
* With memory impairments according to the RL/RI-16 test (free recall≤22 and/or total recall ≤42), according to the thresholds for population-based studies defined by Auriacombe et al., 2010.
* Without memory complaint
* Without dementia Group 3- Cognitively-impaired subjects without dementia and with memory complaints
* MMSE < 24 or < 26 for low and high levels of education, respectively
* With memory impairments according to the RL/RI-16 test (same thresholds as above)
* With memory complaint
* Without dementia

Exclusion Criteria:

* Being left handed
* Presence of dementia (based on the clinical diagnosis)
* Presence of stroke
* Presence of Parkinson's disease
* Presence of a counter-indication for MRI
* Presence of a counter-indication for PET Scan with [18F]-Flutemetamol
* Presence of any health problem preventing travel to the imaging service of the University Hospital
* Being under the legal guardianship of another person or being unable to provide consent to participate
* Pregnant or breastfeeding woman

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Amyloid load | at inclusion (day 0)

SECONDARY OUTCOMES:
Neuropsychological scores | At inclusion (Day 0)
Educational level | At inclusion (Day 0)
Memory complaint | At inclusion (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Michèle ALLARD, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France